CLINICAL TRIAL: NCT00116324
Title: Predicting the Bronchoprotective Response to a Leukotriene Modifier by Genetic Polymorphism
Brief Title: Predicting the Response to Montelukast by Genetic Variation in Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Elliot Israel, MD, Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-P-001696
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Asthma
Keywords: Asthma; Leukotriene receptor antagonist; Hypertonic saline challenge
MeSH Terms: conditions — Asthma | interventions — montelukast

INTERVENTIONS:
Drug: Montelukast

SUMMARY:
The purpose of this study is to examine a specific variation in the genetic code for an enzyme (LTC4 synthase) which plays an important role in the airway inflammation associated with asthma. We hypothesize that asthmatic patients with this variant gene will have a better response to montelukast than patients with the wild type gene, as measured by the ability of montelukast to protect against a hypertonic saline challenge.

DETAILED DESCRIPTION:
Multiple genetic polymorphisms in the leukotriene pathway have been described but their clinical relevance is unclear. A single nucleotide polymorphism in the LTC4 synthase promoter region has been associated with increased LTC4 synthase mRNA and a trend toward improved bronchodilatory response to leukotriene modifiers in severe asthmatics. This study will examine mild to moderate asthmatics with the variant gene and evaluate the bronchoprotective response of montelukast in a double-blind, placebo-controlled cross-over fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 18-55
* Clinical history consistent with asthma
* Mild to moderate asthma as determined by pulmonary function tests--60% or higher of predicted FEV1 for age, sex and race.
* Response to hypertonic saline, which will be the main outcome variable measured.

Exclusion Criteria:

* Smokers (total lifetime smoking history>10 pack-years, any in the past year)
* Pregnant woman-if of childbearing age, not using an acceptable form of birth control.
* Use of a leukotriene modifier within the past month
* Use of inhaled or oral steroids within the past month.
* Emergency room visit for asthma exacerbation within the past 6 weeks.
* Intubation for asthma exacerbation in the past 10 years.
* Adverse reaction to inhaled beta-agonists in the past.
* No recent (past 48 hours) use of anticholinergics, theophylline, antihistamines, pseudoephedrine.
* Patients will also be asked not to use any short acting beta-agonists for 6 hours and long-acting beta-agonists for 48 hours before their initial visit (when pulmonary function evaluation will be performed).
* Lung disease other than asthma
* Significant medical illness other than asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in hypertonic saline PD20

SECONDARY OUTCOMES:
Improved asthma control
Change in exhaled breath condensate inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Drazen JM, O'Brien J, Sparrow D, Weiss ST, Martins MA, Israel E, Fanta CH. Recovery of leukotriene E4 from the urine of patients with airway obstruction. Am Rev Respir Dis. 1992 Jul;146(1):104-8. doi: 10.1164/ajrccm/146.1.104. PMID 1320817
- [Background] Taylor GW, Taylor I, Black P, Maltby NH, Turner N, Fuller RW, Dollery CT. Urinary leukotriene E4 after antigen challenge and in acute asthma and allergic rhinitis. Lancet. 1989 Mar 18;1(8638):584-8. doi: 10.1016/s0140-6736(89)91611-5. PMID 2564113
- [Background] Drazen JM, Yandava CN, Dube L, Szczerback N, Hippensteel R, Pillari A, Israel E, Schork N, Silverman ES, Katz DA, Drajesk J. Pharmacogenetic association between ALOX5 promoter genotype and the response to anti-asthma treatment. Nat Genet. 1999 Jun;22(2):168-70. doi: 10.1038/9680. PMID 10369259
- [Background] In KH, Asano K, Beier D, Grobholz J, Finn PW, Silverman EK, Silverman ES, Collins T, Fischer AR, Keith TP, Serino K, Kim SW, De Sanctis GT, Yandava C, Pillari A, Rubin P, Kemp J, Israel E, Busse W, Ledford D, Murray JJ, Segal A, Tinkleman D, Drazen JM. Naturally occurring mutations in the human 5-lipoxygenase gene promoter that modify transcription factor binding and reporter gene transcription. J Clin Invest. 1997 Mar 1;99(5):1130-7. doi: 10.1172/JCI119241. PMID 9062372
- [Background] Sanak M, Simon HU, Szczeklik A. Leukotriene C4 synthase promoter polymorphism and risk of aspirin-induced asthma. Lancet. 1997 Nov 29;350(9091):1599-600. doi: 10.1016/s0140-6736(05)64015-9. No abstract available. PMID 9393345
- [Background] Sampson AP, Siddiqui S, Buchanan D, Howarth PH, Holgate ST, Holloway JW, Sayers I. Variant LTC(4) synthase allele modifies cysteinyl leukotriene synthesis in eosinophils and predicts clinical response to zafirlukast. Thorax. 2000 Oct;55 Suppl 2(Suppl 2):S28-31. doi: 10.1136/thorax.55.suppl_2.s28. No abstract available. PMID 10992553
- [Background] Anderson PJ, Garshick E, Blanchard JD, Feldman HA, Brain JD. Intersubject variability in particle deposition does not explain variability in responsiveness to methacholine. Am Rev Respir Dis. 1991 Sep;144(3 Pt 1):649-54. doi: 10.1164/ajrccm/144.3_Pt_1.649. PMID 1892306
- [Derived] Kazani S, Sadeh J, Bunga S, Wechsler ME, Israel E. Cysteinyl leukotriene antagonism inhibits bronchoconstriction in response to hypertonic saline inhalation in asthma. Respir Med. 2011 May;105(5):667-73. doi: 10.1016/j.rmed.2010.11.025. Epub 2010 Dec 18. PMID 21169002